CLINICAL TRIAL: NCT03378596
Title: Impact of L-citrulline Associated With L-arginine Supplementation on the Post-exercise Hypotension in Normotensives and Hypertensives
Brief Title: Impact of Citrulline and Arginine Supplementation on the Post-exercise Hypotension (PEH)
Acronym: PEH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Juliano Casonatto (Other)
Responsible Party: Sponsor-Investigator, Juliano Casonatto, Professor, Clinical Research, Universidade Norte do Paraná
Organization: Universidade Norte do Paraná (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-0108
Record Dates: First submitted 2017-12-14; First posted 2017-12-20 (Actual); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Hypertension
Keywords: Post-Exercise Hypotension; Exercise; Arginine; Citrulline
MeSH Terms: conditions — Hypertension; Post-Exercise Hypotension; Motor Activity | interventions — Citrulline; Arginine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- L-citrulline & L-arginine (Experimental): L-citrulline (6 grams) L-arginine (8 grams)
  Interventions: Dietary Supplement: L-citrulline + L-arginine
- L-citrulline & Placebo (Active Comparator): L-citrulline (6 grams) Placebo (6 grams)
  Interventions: Dietary Supplement: L-citrulline; Dietary Supplement: Placebo
- L-arginine & Placebo (Active Comparator): L-arginine (8 grams) Placebo (6 grams)
  Interventions: Dietary Supplement: L-arginine; Dietary Supplement: Placebo
- Placebo (Active Comparator): Placebo (6 grams)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: L-citrulline + L-arginine — L-citrulline + L-arginine - sachet dissolved in water
  Arms: L-citrulline & L-arginine
Dietary Supplement: L-arginine — L-arginine - sachet dissolved in water
  Arms: L-arginine & Placebo
Dietary Supplement: L-citrulline — L-citrulline - sachet dissolved in water
  Arms: L-citrulline & Placebo
Dietary Supplement: Placebo — Placebo (corn starch) - sachet dissolved in water
  Arms: L-arginine & Placebo; L-citrulline & Placebo; Placebo

SUMMARY:
Post-exercise hypotension (PEH) is a established phenomenon as one of the non-pharmacological ways of reducing blood pressure, producing important impacts, particularly in hypertensive individuals. However, the factors involved in the magnitude and duration of this effect are relatively little studied. Thus, the bioavailability of vasodilatation mediators may maximize the duration and magnitude of PEH. In this sense, the objective of the present project will be to verify the impact of L-citrulline associated with L-arginine supplementation on the acute blood pressure response after an aerobic exercise session. Approximately 80 adults (40 normotensive and 40 hypertensive) will be selected. The sample will be submitted to measurements of body mass, height and resting blood pressure. After the minimum interval of 48 h, subjects will be randomly submitted to four experimental situations (exercise/L-citrulline, exercise/L-arginine, exercise/placebo, exercise/L-citrulline + L-arginine). The exercise sessions (40 min in treadmill at 60% of FCres) will be performed with a minimum interval of 48 h. After each session, the blood pressure of the sample will be recorded during 24 hours. For data analysis, blood pressure values will be plotted in average of the wakefulness and average of the sleep periods and average of the 24 hours. The comparisons will be made through the ANOVA (repeated measures), following the recommended assumptions. It is hoped that the results of this project will collaborate to the knowledge regarding non-pharmacological models aimed at the prevention and treatment of hypertension in normotensive and hypertensive patients.

DETAILED DESCRIPTION:
Participants After sample size calculation (see statistical analysis session), 40 hypertensives and 40 normotensive sedentaries will be recruited to this study. All volunteers (both sexes) will be adults without osteoarticular disabilities and they will need a medical authorization to physical exercise practice. Participants will be recruited from an exercise program project linked to the university that offered stretching and functional exercises sessions to the external community. The study follow the Declaration of Helsinki and the Institutional Ethics Committee approved all experimental procedures and protocols. Each participant will be fully informed of all potential risks and experimental procedures, after which, informed written consent will be signed. Table 1 shows the basics characteristics of the participants.

Study design A double-blind crossover randomized clinical trial will be conducted. After the minimum interval (48 hours), the subjects will be randomly (using a random number table - https://www.random.org/) submitted to four experimental situations (exercise/L-citrulline, exercise/L-arginine, exercise/placebo, exercise/L-citrulline + L-arginine). The participants will ingested a sachet, which contained L-citrulline malate (6 grams) or L-arginine (8 grams) or placebo (6 grams of corn starch) dissolved in water.

The substances will be ingested 120 minutes before the experimental or control session. Anthropometric measures will be taken before the rest period. The exercise session consisted of 5 min to warm up (50% of 65% HRreserve) and 40 minutes of run/walk at 60-70% HRreserve (or 12-14 ratings of perceived exertion [RPE](1) if take some beta-blocker medicines) in a treadmill. This will be followed by a progressive cooldown (5 minutes). In the control session, the participants will be remained seated in a quiet room for 40 min.

After the exercise/control sessions, the blood pressure will be measured every 10 minutes over the course of 60 minutes and the heart rate variability will be recorded continuously for 60 minutes (laboratorial phase). Then, 15 minutes will be given to the participants to take a shower and change the clothes before the ambulatory blood pressure device be attached on their arm. The ambulatory blood pressure will be recorded over 24 hours. In the next day, the participants will be asked to return to the laboratory to remove the device.

Anthropometry The weight will be measured by the digital anthropometric scale (Urano, OS 180A, Canoas, Brasil), with accuracy of 0.1kg and height will be measured by stadiometer with accuracy of 0.1cm, in accordance with the procedures described by Gordon et al (2). The body mass index (BMI) will be defined as the body mass (kg) divided by the square of the body height.

Office Blood Pressure (laboratorial phase) The office blood pressure measurements will be taken with oscillometric device (Omron MX3 Plus, Bannockburn, EUA) previously validated for clinic measures in adults (3). Firstly, the participants remained seated (rest period) in calm, quiet and thermoneutral (22°-24°C) environment for 20 min. The blood pressure will be measured three times during the rest period (at 10 min, 15 min and 20 min). The rest blood pressure value will be considered as the average of these three measurements. Immediately following the sessions (exercise or control), the blood pressure will be measured in a quiet environment during 60 minutes. The blood pressure measurements will be taken according to the American Heart Association recommendations (4).

Heart rate variability measures The heart rate variability will be monitored during the rest period using a cardiac monitor (Polar RS800CX, Kempele, Finlândia) previously validated (5). The recorded R-R intervals will be transferred to a computer using a specific software (Polar Pro-Trainer software, Kempele, Finlândia). The Fast Fourier Transformation will be applied to quantify the low and high frequencies in to normalized units, in accordance with Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology (6). The participants will be taking beta-blockers will be excluded of this analysis.

The time domain analisys will be obtained by SDNN (standard deviation of the NN interval), RMSSD (the square root of the mean of the sum of the squares of differences between adjacent NN intervals), pNN50 (NN50 count divided by the total number of all NN intervals), indexes. The range interval analysis will be 5 min (rest, previous exercise) and 30 min (post-exercise - laboratorial phase) using the Kubios HRV, version 2.2 (Kuopio, Finlândia).

Ambulatorial blood pressure measures (ambulatorial phase) The ambulatorial blood pressure measurements will be taken with oscillometric device (Dyna-MAPA - São Paulo, Brazil) attached on the left arm, always by the same investigator, in accordance with procedures described by American Heart Association (4). The participants will be instructioned to keep the arm stand during the measures. The device will be calibrated by direct comparison with mercury sphygmomanometer, by trained technical person, in agreement with recommendations (4).

The monitor will be setting to register the systolic and diastolic blood pressure and heart rate every 20 minutes during "daytime" (08:00am to 11:00pm) and every 30 minutes during "night-time" (11:00pm to 08:00am) to reduce sleep disturbs. The device screen will be electronically blinded to avoid feedback. All participants will be instructed to register and reported their sleep time in a diary on the day after.

The data will be recorded in the device memory, then they will be send to a computer using specific software (Aplicação Dyna Mapa - Version 5.0.382.12) for analysis. The average of the valid readings will be above 90% for all participants.

Statistical analysis Assuming a standard deviation of 5 mmHg(7) for the systolic blood pressure, an alpha of 5% and a desired statistical power of 80% for detecting a minimum difference of 7 mmHg (7) required 10 subjects in each group.

The datas will be presented in the text as mean and standard error. The sphericity Mauchly´s test will be applied. Greenhouse-Geisser correction will be used if necessary. Then, these datas will be compared with a one-factor repeated measures general linear model (GLM). Fisher multiple comparisons will be employed to examine differences between pairs of trials.

The ambulatory blood pressure will be analysed as awake, sleep and 24 hours of monitoring. Statistical significance will be defined as P<0.05. The statistical analysis will be generated using SPSS, version 20, system for windows.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive and Normotensive, without osteoarticular disabilities and medical authorization to physical exercise practice.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-01-02 (Estimated); Primary Completion 2018-01-31 (Estimated); Study Completion 2018-02-28 (Estimated)

PRIMARY OUTCOMES:
Ambulatorial Blood Pressure Monitoring | 24 hours
  The ambulatorial blood pressure measurements will be taken with oscillometric device (Dyna-MAPA - São Paulo, Brazil) attached on the left arm. The participants will received instructions to keep the arm stand during the measures. The monitor will be setting to register the systolic and diastolic blood pressure and heart rate every 20 minutes during "daytime" (08:00am to 11:00pm) and every 30 minutes during "night-time" (11:00pm to 08:00am) to reduce sleep disturbs. The device screen will be electronically blinded to avoid feedback. The metric measures will be reported by millimeters of mercury (mmHg).

CONTACTS AND LOCATIONS:
Locations (1):
- Juliano Casonatto, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Borg G. Borg's Perceived Exertion and Pain Scales. Champaign: Human Kinetics; 1998.
- [Background] Gordon CC, Chumlea WC, Roche AF. Stature, recumbent length, and weight. Lohman TG, Roche AF, Martorell R, editors. Champaign: Human Kinetics Books; 1988. 3-8 p.
- [Background] Coleman A, Freeman P, Steel S, Shennan A. Validation of the Omron MX3 Plus oscillometric blood pressure monitoring device according to the European Society of Hypertension international protocol. Blood Press Monit. 2005 Jun;10(3):165-8. doi: 10.1097/00126097-200506000-00009. PMID 15923819
- [Background] Pickering TG, Hall JE, Appel LJ, Falkner BE, Graves J, Hill MN, Jones DW, Kurtz T, Sheps SG, Roccella EJ; Subcommittee of Professional and Public Education of the American Heart Association Council on High Blood Pressure Research. Recommendations for blood pressure measurement in humans and experimental animals: Part 1: blood pressure measurement in humans: a statement for professionals from the Subcommittee of Professional and Public Education of the American Heart Association Council on High Blood Pressure Research. Hypertension. 2005 Jan;45(1):142-61. doi: 10.1161/01.HYP.0000150859.47929.8e. Epub 2004 Dec 20. PMID 15611362
- [Background] Quintana DS, Heathers JA, Kemp AH. On the validity of using the Polar RS800 heart rate monitor for heart rate variability research. Eur J Appl Physiol. 2012 Dec;112(12):4179-80. doi: 10.1007/s00421-012-2453-2. Epub 2012 Jul 13. No abstract available. PMID 22790488
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Casonatto J, Tinucci T, Dourado AC, Polito M. Cardiovascular and autonomic responses after exercise sessions with different intensities and durations. Clinics (Sao Paulo). 2011;66(3):453-8. doi: 10.1590/s1807-59322011000300016. PMID 21552672
- [Derived] Domingues V, Cavalari JV, Grandolfi K, Aguiar AF, Borghi SM, Casonatto J. Acute Effects of Citrulline Malate Supplementation on Nocturnal Blood Pressure Dipping After Exercise in Hypertensive Patients: A Randomized, Placebo-Controlled Trial. J Diet Suppl. 2024;21(6):868-880. doi: 10.1080/19390211.2024.2414052. Epub 2024 Oct 10. PMID 39385595